CLINICAL TRIAL: NCT05061355
Title: Antibiotics Vs Antibiotics and Surgical ThERapy for Infective Endocarditis
Acronym: ASTERIx
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Emil Loldrup Fosbol (Other)
Collaborators: Herlev and Gentofte Hospital (Other); Bispebjerg Hospital (Other); Amager Hospital (Other); Nordsjaellands Hospital (Other); Copenhagen University Hospital, Hvidovre (Other)
Responsible Party: Sponsor-Investigator, Emil Loldrup Fosbol, MD, PhD, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-21014406
Record Dates: First submitted 2021-09-08; First posted 2021-09-29 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-04

CONDITIONS: Endocarditis Infective
Keywords: Surgery; Medical care
MeSH Terms: conditions — Endocarditis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Surgery plus medical therapy (Experimental): Heart valve surgery will be performed as soon as possible and preferably within 48 hours of randomization in addition to standard medical care for IE.
  Interventions: Procedure: Heart valve surgery
- Medical therapy (No Intervention): Only standard medical care for IE.

INTERVENTIONS:
Procedure: Heart valve surgery — Heart valve surgery will be performed as soon as possible and preferably within 48 hours
  Arms: Surgery plus medical therapy

SUMMARY:
Infective endocarditis (IE) is a deadly disease and the incidence is increasing. An important initial assessment of patients with IE includes whether surgical treatment is indicated; yet, appropriate data to guide this assessment do not exist.

The ASTERIx study will assess whether a surgical approach in addition to medical care for treatment of IE is superior to medical care alone. In total, 496 patients will be included in the study over four years. The study is event-driven and will require at least 240 events. The study will assess the primary composite outcome of death, embolization, relapse of IE, new heart failure or reinfection.

Study participants who survive to discharge will be followed by routine clinical check-ups at one- and four-weeks post-discharge and at three months. Additionally a 12-month study follow-up is planned.

The investigators will also conduct a small substudy to assess the frequency of silent emboli.

DETAILED DESCRIPTION:
Infective endocarditis (IE) is a life-threatening disease and studies suggest that the incidence of IE has almost doubled in the last twenty years. Despite improved disease-management and diagnostics (i.e. antibiotics, surgery, and imaging techniques) IE remains a condition that is hard to diagnose and associated with high mortality (≈1/3 die within one year). Surgery is a key part of the clinical practice in IE, but the role of surgery has been greatly debated and is also used with great variation among centers. Valve repair and replacement are high-risk procedures and per-operative risk is therefore also a natural part of decision for surgery. Clinical guidelines on surgical indications have remained stable in the past decades; however, these recommendations are not based on randomized data and at the moment we are putting very sick patients with endocarditis through high-risk procedures without the proper knowledge and perhaps we refrain from surgery where benefit may be likely.

Eligible patients for study inclusion (inclusion criteria are met), will be assessed at the respective departments in Denmark where IE patients are treated (or in similar department for the international centers). All departments refer to a local endocarditis heart team at a tertiary center with cardiothoracic surgical capabilities. If no exclusion criteria exist (confirmed by the local endocarditis heart team) and the patients sign informed consent after a decent time for reflection (24 hours) then randomization will be done as soon as possible. Study participants with IE are randomized to either:

1. Medical Therapy and surgery: Standard of care treatment with antibiotics according to national and international guidelines depending on the microbiological agent and the investigators aim to perform surgery within 48 hours of randomization.
2. Medical Therapy alone with standard of care treatment with antibiotics according to guidelines depending on the microbiological agent.

Point of randomization will be in the hospital when the patient is assessed for open heart valve surgery by the heart team.

If study participants are included in the study and are randomized to the medical treatment arm of the trial, participants will stay at the local IE center and continue treatment there. If participants are randomized to surgery, the participants will be transferred to a tertiary center as soon as possible and returned to the non-surgical center for completement of treatment. After end of treatment all participants will be discharged to routinely follow-up at one- and four-weeks and at three months. Additionally, a 12 months visit will be planned for all study participants.

ELIGIBILITY:
Inclusion Criteria:

Definite left-sided infective endocarditis defined by the ESC (European Society of Cardiology) modified Duke Criteria

AND

Valve vegetation =>10mm AND <=30mm with 1 or no previous embolic event during current IE case

Exclusion Criteria:

* Unwilling to sign informed consent
* At least one clear class I recommendation for surgery because of heart failure or uncontrolled local infection (abscess, false aneurysm, fistula)
* Unavailable for follow-up (e.g. tourist)

OR

At least one of the following criteria (unsuitable for surgery)

* Intracranial hemorrhage <1 month
* Life expectancy <1 year
* Age ≥85 years
* BMI below 15 or above 45
* Possible severe liver cirrhosis (Child-Pugh Class B or worse)
* Clinical frailty score of 5 or above
* EUROSCORE II > 50%
* Severe pulmonary disease (FEV1 (Forced expiratory volume in 1 second) or DLCO (Diffusing capacity for carbon monoxide) <30% of expected)
* Left ventricular ejection fraction (<20%)
* Technically inoperable (e.g. extracorporeal circulation deemed impossible)

Ages: 18 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 496 (Estimated)
Dates: Start 2021-09-09 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality (Death) among study participants after randomization | It will be assessed at discharge, and every year thereafter
  The incidence of all-cause mortality will be compared between treatment groups (medical therapy vs. medical therapy + surgery). [Date on all-mortality will be assessed in the ASTERIx study database REDCap (electronic Case Report File (eCRF)) and all information in the database are gathered from the study participants medical records].
Number of study participants with clinical stroke (persisting symptoms >24 hours from onset) after randomization | It will be assessed at discharge, and every year thereafter
  The incidence of stroke with corresponding clinical signs of stroke (e.g., sudden numbness or weakness of the face, arm or leg, typically in one side of the body, confusion: trouble speaking or understanding speech etc.). [The information on clinical stroke are assessed in the study participants medical records which contains information on imaging modalities and this information are entered in the ASTERIx REDCap database. ]
Number of study participants with systemic embolization after randomization | It will be assessed at discharge, and every year thereafter
  New embolic event (with corresponding symptoms from the affected organ/organs), to one of the following organs:
  * Brain
  * Kidney
  * Spleen
  * Eyes or
  * Extremities
  [Information on embolic events are gathered from study participants medical records which includes imaging modalities e.g., PET-CT. Information on new embolic events will be entered in ASTERIx REDCap database, only date of first embolic event after randomization are entered into REDCap.]
Number of study participants with new endocarditis event after randomization | It will be assessed at discharge, and every year thereafter
  The incidence of new endocarditis event after randomization are defined as followed:
  * Relapse of bacteria with the same organism > 7 days after study intervention
  * Vegetation enlargement (>50%) or local spreading of infection assessed by echocardiography .
  * Re-infection after complete treatment for the initial endocarditis episode.
  [All the listed outcomes defining new endocarditis event will be assessed from study participants medical records including information from the Danish Microbiology Database and entered into ASTERIx REDCap database]
Number of study participants hospitalized for Heart Failure (HF) after randomization | It will be assessed at discharge, and every year thereafter
  The incidence of hospitalization for Heart Failure among study participants. [Information are gathered from medical records and entered into ASTERIx REDCap database].

SECONDARY OUTCOMES:
Individual components of the primary endpoint at study conclusion | It will be assessed at discharge, and every year thereafter
  One of the 5 individual components of the composite primary outcome. [Please see detailed description in the description of each individual component of the primary outcome].
Number of study participants undergoing unplanned heart valve surgery due to IE after randomization | It will be assessed at discharge, and every year thereafter
  Incidence of unplanned heart valve surgery due to IE. [Information gathered from medical records and entered into ASTERIx REDCap database].
Number of study participants with end-stage renal disease and in need of renal replacement therapy after randomization | It will be assessed at discharge, and every year thereafter
  Incidence of renal replacement therapy (RRT) among study participants WITHOUT RRT prior to date of randomization. [Information regarding RRT will be gathered from study participants medical records and entered in ASTERIx REDCap database].
Number of study participants with either implantation of a Pacemaker or Pacemaker extraction after randomization. | It will be assessed at discharge, and every year thereafter
  The incidence of pacemaker implantations and extractions among study participants. [Information on Pacemaker implantation or extraction will be gathered from study participants medical records and entered into ASTERIx REDCap database]
Cause-specific mortality (Death) among study participants after randomization. | It will be assessed at discharge, and every year thereafter
  Incidence of cause-specific mortality (See definition below)
  Definition of cause-specific mortality:
  * Cardiovascular OR
  * Non-cardiovascular (infectious, malignancy, other, and unknown)
  [Date will gathered from medical records and entered into ASTERIx REDCap database].
Number of days in hospital. | It will be assessed at discharge, and every year thereafter
  Length of stay in hospital among study participants will be defined as:
  1. From date of admission until date of discharge
  2. From date of randomization until date of discharge [Date will be gathered from study participants medical records and entered into ASTERIx REDCap date. The actual number of dates will be calculated as followed {date of discharge} - {date of admission/date of randomization}]
Clinical status at discharge | It will be assessed at discharge, and every year thereafter
  Composite outcome measuring the incidence of:
  * need for help with daily activities
  * use of utilities for walking,
  * home help
  * discharged to nursing facility or
  * disability pension [Date will be gathered from medical records and entered into ASTERIx REDCap database. Information on disability pension will be received through register-linkage].

OTHER OUTCOMES:
Number of study participants suffering from silent embolic event (without any clinical symptoms) after randomization | It will be assessed at point of randomization and 4 weeks after
  To assess frequency of silent emboli, we perform magnetic resonance imaging of the brain on day of randomization and 4 weeks after. A total of 60 patients (30 patients in each arm) will be included in this substudy. This small substudy will be conducted at Copenhagen University Hospital (Rigshospitalet)

CONTACTS AND LOCATIONS:
Overall Officials: Emil L Fosbol, MD, Ph.D, Principal Investigator — Rigshospitalet, Denmark
Locations (15):
- Denmark (9):
  - Aalborg University Hospital, Aalborg
  - Aarhus University Hospital, Aarhus
  - University Hospital of Copenhagen, Rigshospitalet, Copenhagen
  - Amager Hvidovre Hospital, Copenhagen
  - Bispebjerg Hospital, Copenhagen
  - Herlev and Gentofte Hospital, Gentofte Municipality
  - Nordsjællands Hospital, Hillerød
  - Odense University Hospital, Odense
  - Zealand University Hospital, Roskilde
- Leipzig Heart Center, Leipzig, Germany
- Netherlands (3):
  - Amsterdam University Medical Center, Amsterdam
  - Catharina Hospital, Eindhoven
  - Leiden University Medical Center, Leiden
- Sweden (2):
  - Karolinska Institutet, Stockholm, Solna
  - Linköping Heart Center, University Hospital, Linköping

IPD SHARING:
Plan to Share IPD: No